CLINICAL TRIAL: NCT05015127
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2/3 Operational Seamless Design Clinical Study to Evaluate the Efficacy and Safety of HBM9161 Subcutaneous Injection in Chinese Patients With Active, Moderate to Severe Thyroid Eye Disease (TED)
Brief Title: A Study to Evaluate the Efficacy and Safety of HBM9161 on Moderate to Severe Thyroid Eye Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9161.5
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-11

CONDITIONS: Thyroid Ophthalmopathy
Keywords: TED
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — HBM9161

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- HBM9161 680 mg qw by q2w from week 13 (Experimental): Subcutaneous injection; HBM9161 680 mg qw from week 13
  Interventions: Drug: HBM9161 680 mg qw by q2w from week 13
- HBM9161 680 mg qw by q2w from week 7 (Experimental): Subcutaneous injection; HBM9161 680 mg qw by q2w from week 7
  Interventions: Drug: HBM9161 680 mg qw by q2w from week 7
- Placebo (Experimental): Subcutaneous injection; Placebo
  Interventions: Drug: Placebo
- Placebo qw by HBM9161 680mg qw from week 12 (Experimental): Placebo qw by HBM9161 680mg qw from week 12
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HBM9161 680 mg qw by q2w from week 13 — HBM9161 680 mg qw by q2w from week 13
  Arms: HBM9161 680 mg qw by q2w from week 13
Drug: Placebo — Placebo
  Arms: Placebo
Drug: HBM9161 680 mg qw by q2w from week 7 — HBM9161 680 mg qw by q2w from week 7
  Arms: HBM9161 680 mg qw by q2w from week 7
Drug: Placebo — Placebo qw by HBM9161 680mg qw from week 12
  Arms: Placebo qw by HBM9161 680mg qw from week 12

SUMMARY:
Primary Objective: To preliminarily evaluate the efficacy of the treatment regimen of HBM9161 680 mg administered subcutaneously weekly and sequentially every other week for 12 weeks in Chinese patients with active moderate to severe TED.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind and placebo-controlled study. The investigational drug is HBM9161 injection, with the indication of TED. Subjects will be randomized to treatment group I, treatment group II, or placebo group. Subjects in treatment group 1 will receive HBM9161 680 mg subcutaneously once weekly (qw) for 12 doses; Subjects in treatment group 2 will receive HBM9161 680 mg subcutaneously once weekly (qw) for 6 doses, followed by HBM9161 680 mg subcutaneously once every two weeks (q2w) for 3 doses; Subjects in placebo group will receive placebo subcutaneously once weekly (qw) for 12 doses. After the 12-week dosing period, there will be a 5-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent form.
2. Male or female between the ages of 18 and 70 (including boundary values).
3. Active TED associated with a clinical diagnosis of Graves' disease or Hashimoto's thyroiditis with CAS ≥ 3 at the screening visit and baseline (both on a 7-item scale) in the eye with the most severe proptosis.
4. The active period of TED starts within 9 months prior to screening visit
5. Positive anti-TSHR antibody at screening visit.
6. Subject is willing and able to receive treatment and complete corresponding assessments as required by the protocol.

Exclusion Criteria:

1. Other uncontrolled concurrent diseases
2. Serious TED requiring surgery or radiotherapy
3. Suffer from autoimmune diseases or ophthalmic conditions other than TED that, in the opinion of the investigator, would impact the assessment of the study drug
4. No significant laboratory abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proptosis responder rates of the treatment groups and placebo group at Week 12 | At week 12
  Proptosis responder rates of the treatment groups and placebo group at Week 12

SECONDARY OUTCOMES:
The percentage of subjects with a CAS value of 0 or 1 in the study eye | At week 6, week 12, week 18 and week 24
  The percentage of subjects with a CAS value of 0 or 1 in the study eye
The change from Baseline in proptosis measurement in the study eye | At week 6, week 12, week 18 and week 24
  The change from Baseline in proptosis measurement in the study eye
Composite responder rate | At week 6, week 12, week 18 and week 24
  Composite responder rate
Diplopia response rate | At week 6, week 12, week 18 and week 24
  Diplopia response rate
The change from baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire visual function score and psychosocial function score | At week 6, week 12, week 18 and week 24
  The change from baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire visual function score and psychosocial function score
The changes in proptosis responder rate over time | From week 1 to week 24
  The changes in proptosis responder rate over time
The change from baseline in quantitative measurement of orbital structures by MRI, including exophthalmos values, fatty tissue thickness of inner side in eye balls, thickness of extraocular muscles. All the above parameters will be measured in millimeter | At week 12, week 24
  The change from baseline in quantitative measurement of orbital structures by MRI, including exophthalmos values, fatty tissue thickness of inner side in eye balls, thickness of extraocular muscles. All the above parameters will be measured in millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Zhou, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No